CLINICAL TRIAL: NCT00303004
Title: Combination Treatment With Bosentan and Sildenafil to Patients With Eisenmengers Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Kasper Iversen, Rigshospitaler
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 01000
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2008-01-24 (Estimated); Status verified 2008-01

CONDITIONS: Eisenmenger Syndrome
MeSH Terms: conditions — Eisenmenger Complex | interventions — Bosentan; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bosentan and Sildenafil

SUMMARY:
The purpose of this study is to investigate if combination treatment with Bosentan and Sildenafil to patients with Eisenmenger syndrome is beneficial.

DETAILED DESCRIPTION:
Eisenmengers syndrome is condition with severe pulmonary arterial hypertension due to a shunting of blood from the left side of the heart to the right side of the heart. When the pressure in the pulmonary arteries levels the systemic blood pressure, blood begins to shunt from the right side of the heart to the left side of the heart leading to a condition with cyanosis, impaired physical capacity and increased mortality (Eisenmengers syndrome).

Several clinical trials have shown that there is a beneficial effect of treating patients with primary pulmonary arterial hypertension with Bosentan or Sildenafil and that a combination of these may have an additive or even synergistic effect. No clinical trials with Sildenafil and Bosentan has been conducted for patients with Eisenmengers syndrome. Observational studies and case stories indicate however that the effect of Bosentan or Sildenafil in patients with Eisenmengers syndrome may be as promising in these patients as in patients with primary pulmonary arterial hypertension.

We would like to examine the effect of treating patients with Eisenmengers Syndrome with a combination of Bosentan and Sildenafil.

The primary end point is change in physical performance measured with six minutes walking test.

Secondary end points is change in saturation, NYHA class, cardiac output (cardiac catheterization and innocor measurement), pulmonary vascular resistance (cardiac catheterization) shunt ratio (MRI), strain of right ventricle (BNP and echocardiography), quality of life and serum erythropoitin.

The trial is designed as a randomized, single centre, placebo controlled, double blind cross over study.

Twenty patients with Eisenmengers syndrome is included. All patients will be treated in three months with Bosentan. There after patients will be randomized to receive either Sildenafil (50 mg tid) or placebo as add on therapy for three month. Hereafter a cross over will be made and patients in combination treatment will receive only their native treatment and vice versa.

Examinations for primary and secondary endpoints will be made at baseline, before cross over and at the end of the study. All up titrating of medication will be performed during admittance. Patients will during the study period be close monitored with registration of adverse advents, physical examination and blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Eisenmenger syndrome
* Negative pregnancy test

Exclusion Criteria:

* Elevated liver enzymes to more than 3´times normal value
* Hypotension (SBP < 90 mmhg).
* Mandatory treatment with nitrates
* Myocardial infarction within 3 months
* Stroke within 3 months
* Known allergy to Bosentan or Sildenafil
* inherited degenerative diseases in retina
* Breast feeding
* Suspicion of risc of noncompliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
6 minutes walking distance

SECONDARY OUTCOMES:
Pulmonary blood flow
Systemic blood flow
Pulmonary resistance
Shunt ratio
Erythropoitin
BNP
Saturation in rest
Saturation in activity
Quality of life
Right ventricle systolic and diastolic function
Working capacity
Oxygen consumption at rest
Oxygen consumption during maximal work

CONTACTS AND LOCATIONS:
Overall Officials: Lars Soendergaard, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Iversen K, Jensen AS, Jensen TV, Vejlstrup NG, Sondergaard L. Combination therapy with bosentan and sildenafil in Eisenmenger syndrome: a randomized, placebo-controlled, double-blinded trial. Eur Heart J. 2010 May;31(9):1124-31. doi: 10.1093/eurheartj/ehq011. Epub 2010 Mar 3. PMID 20202971